CLINICAL TRIAL: NCT03068832
Title: A Pilot Study to Assess the Safety, Feasibility, and Preliminary Efficacy of a Neoepitope-based Personalized Vaccine Approach in Pediatric Patients With Recurrent Brain Tumors
Brief Title: Neoepitope-based Personalized Vaccine Approach in Pediatric Patients With Recurrent Brain Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Made the decision to not go forward with the study
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201807123
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Pediatric Brain Tumor
MeSH Terms: interventions — poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Personalized peptide vaccine and poly-ICLC (Experimental): * The synthetic long peptide(s) and poly-ICLC will be given on Cycle 1 Day 1 when available.
  * Additional peptide vaccine doses will be administered again on Days 4, 8, 15, and 22 of the first cycle as a priming strategy. On all subsequent cycles, the peptide vaccine will be given on Day 1.
  * Peptide vaccine administration will continue until supply is exhausted or development of intolerance or disease progression in the case of fatal high grade neoplasms. Otherwise, vaccination will continue until supply is exhausted or intolerance or one year for non-fatal tumors. Additionally, patients with non-fatal tumors who complete one year of vaccinations and have stable disease will be given the option of resuming vaccinations if they develop subsequent progression if remaining vaccine is available.
  Interventions: Biological: Personalized peptide vaccine; Drug: Poly ICLC; Procedure: Peripheral blood draw

INTERVENTIONS:
Biological: Personalized peptide vaccine — -It may take 3-4 months for sequencing, neoantigen prediction, and peptide manufacturing
Drug: Poly ICLC — -Poly-ICLC is supplied by Oncovir in single-dose vials containing 1 mL of 2 mg/mL opalescent white suspension.
  Other Names: Poly-ICLC; Hiltonol
Procedure: Peripheral blood draw — * After trial enrollment and up to 7 days after the 1st vaccine dose
  * 2 weeks after last dose
  * Time of progression or discontinuation

SUMMARY:
The early clinical development paradigm for chemotherapeutic agents has significantly influenced the development of therapeutic cancer vaccines. However, there are major differences between these two classes of therapeutics that have important implications for early clinical development. Specifically, the phase 1 concept of dose escalation to find a maximum-tolerated dose does not apply to most therapeutic cancer vaccines. Most therapeutic cancer vaccines are associated with minimal toxicity at a range that is feasible to manufacture or administer, and there is little reason to believe that the maximum-tolerated dose is the most effective dose.

In a recent article from the biostatistics literature, Simon et al. write that "the initial clinical trial of many new vaccines will not be a toxicity or dose-ranging trial but rather will involve administration of a fixed dose of vaccine … in most cases the dose selected will be based on preclinical findings or practical considerations. Using several dose levels in the initial study to find the minimal active dose or to characterize the dose-activity relationship is generally not realistic".

Consistent with these recommendations, the general philosophy of the phase 1 clinical trial is to facilitate a prompt preliminary evaluation of the safety and immunogenicity of the personalized synthetic long peptide vaccine strategy. The proposed clinical trial will test a fixed dose of vaccine. There is considerable experience with the synthetic long peptide vaccine platform. The synthetic long peptide vaccine platform has an excellent safety profile, and the optimal dose appears to be based on practical considerations (solubility of the peptide). The dose to be tested in the proposed clinical trial is consistent with other similar cancer vaccine trials that have been recently completed or are currently ongoing. The sample size (n=10-20) will provide a reasonably reliable estimate of the safety and immunogenicity of the vaccine.

ELIGIBILITY:
It is anticipated that most potential participants will be consented following standard of care surgical procedure (biopsy, resection). Consenting and eligible patients will have sequencing data accessed to evaluate for candidate neoantigens (sequencing may take place under the auspices of this project, as part of the participant's standard of care, or under a tumor bank or other research project). Shortly before the vaccine is ready for administration, participants will be re-screened using the criteria below to confirm eligibility.

Inclusion Criteria:

* Any patient, regardless of current age, who was diagnosed between the ages of 0-21 years with a pediatric brain tumor of any histologic subtype, who has now developed recurrent or refractory disease.
* Availability of tissue for sequencing to determine presence of targetable neoantigen. This may be fresh tissue collected as part of routine care, another research project or archived tissue from a previous craniotomy with biopsy, subtotal resection, total gross resection, or re-resection.
* Karnofsky/Lansky performance status ≥ 60%
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (IULN)
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine ≤ IULN OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Systemic corticosteroid therapy is permitted provided dosing is minimal based on age 0.1mg/kg/day with a max of 4mg daily (dexamethasone or equivalent) on the day of vaccine administration.
* Bevacizumab will be allowed if given for symptomatic control of vasogenic edema and to avoid high dose of corticosteroids at the discretion of the treating physician.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* As this is a safety and feasibility study, prior immunotherapy will be permitted. However, any prior immunotherapy must be discontinued at least 2 weeks before peptide vaccine administration. Non-immunologic therapy may be continued.
* No candidate neoantigen identified during screening.
* A history of other malignancy ≤ 3 years previous with the exception of non-melanoma skin cancer, any in situ cancer that has been successfully resected and cured, treated superficial bladder cancer, or any early-stage solid tumor that was successfully resected without need for adjuvant radiation or chemotherapy.
* Currently receiving any other investigational agents.
* Known allergy, or history of serious adverse reaction to, vaccines such as anaphylaxis, hives, or respiratory difficulty.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to poly-ICLC or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of pre-existing immunodeficiency disorder, autoimmune condition requiring immunosuppressive therapy, or chronic infection (i.e. hepatitis B, hepatitis C, HIV). This includes inflammatory bowel disease, ulcerative colitis, Crohn's disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjögren's syndrome, sarcoidosis, or other rheumatologic disease or any other medical condition or use of medication which might make it difficult for the patient to complete the full course of treatments or to generate an immune response to vaccines.
* Presence of clinically significant increased intracranial pressure (e.g. impending herniation) or hemorrhage, uncontrolled seizures, or requirement for immediate palliative treatment.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 7 days of first dose of vaccine.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-30 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of adjuvant personalized neoantigen peptide vaccine administration with poly-ICLC as measured by grade 3 and 4 adverse events | Up to 30 days following last day of study treatment (up to 4 months)
  -As defined by CTCAE v. 4.03
Feasibility of adjuvant personalized neoantigen peptide vaccine administration with poly-ICLC as measured by the number of participants who have a neoantigen specific long peptide vaccine identified and generated | 12-14 weeks
  -The vaccine study drug is a frozen solution for injection. It is a personalized vaccine composed of up to 20 synthesized peptides that are approximately 20 to 35 amino acids in length. The peptides are designed to generate an immune response to neoantigens found in each patient's tumor.

SECONDARY OUTCOMES:
Characterize tumor-infiltrating lymphocytes (TIL) | Up to 2 weeks after the last dose (up to 4 months)
  -Paired t-test or paired-sample Wilcoxon Signed Rank test will be used to compare the gene expression of TIL in blood as measured before and after treatment.
Frequency of expressed neoantigens using patient-specific HLA class I prediction algorithms | Completion of treatment (up to 3 months)
  -Up to 20 of the highest priority sequencing-identified mutant tumor-specific antigens that are confirmed to bind and stabilize HLA class I molecules will be targeted

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Rubin, M.D., Ph.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu